CLINICAL TRIAL: NCT02283255
Title: Cardiovascular, Pulmonary and Skeletal Muscle Evaluation in Patients With Univentricular Physiology in the Late Postoperative Period of the Fontan Surgery: Effects of Exercise Training
Brief Title: Cardiovascular, Pulmonary and Skeletal Muscle Evaluation Postoperative in Fontan Patients: Effects of Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Aida Luiza R Turquetto, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 01998712.7.0000.0068
Record Dates: First submitted 2014-09-03; First posted 2014-11-05 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Congenital Heart Disease; Single Ventricle; Univentricular Heart
Keywords: Fontan; Exercise; Pulmonary Function; Aerobic Capacity; Skeletal Muscle; Neurovascular control; Functional capacity
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart; Motor Activity | interventions — beta-Aminoethyl Isothiourea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Training Group (Active Comparator): Aerobic Training: Aerobic training and muscle strength exercise for upper and lower limbs, 3 times a week for 4 months.
  Interventions: Other: Aerobic Exercise Training
- Inspiratory Muscle Training Group (Active Comparator): Respiratory Training: muscle training using POWERbreathe device, 7 times a week, 3 series of 30 repetitions per day, for 4 months.
  Interventions: Other: Inspiratory Muscle Training
- No Exercise Trainint Group (Active Comparator): No Physical Activity: Control group (usual care)
  Interventions: Other: No Exercise Training

INTERVENTIONS:
Other: Aerobic Exercise Training — Supervised aerobic and light muscle resistance exercise training
  Other Names: AET
  Arms: Aerobic Exercise Training Group
Other: Inspiratory Muscle Training — Inspiratory muscle training with POWERbreathe device
  Other Names: IMT
  Arms: Inspiratory Muscle Training Group
Other: No Exercise Training — Usual care
  Other Names: NET
  Arms: No Exercise Trainint Group

SUMMARY:
Introduction: The Fontan operation is the surgical treatment in most patients with either anatomic or functional single ventricles. In this operation, the subpulmonary ventricle is bypassed, connecting the systemic veins directly to the pulmonary arteries. The lack of a subpulmonary ventricle is associated with a nonpulsatile pulmonary flow and triggers a sequence of adaptive mechanisms along the life of these patients. The most frequent consequence of these adaptative mechanisms is the reduction in functional capacity, objectively measured by the decrease in peak oxygen consumption (VO2). So, cardiovascular and pulmonary functioning and skeletal muscle alterations can explain exercise intolerance in these patients.

Objectives: 1. To compare the cardiovascular, pulmonary, and musculoskeletal system variables in clinically stable Fontan patients with Healthy subjects; 2. To correlate the variables of the cardiovascular, pulmonary, and skeletal muscle with the functional capacity in Fontan patients; 3. To identify predictors of low functional capacity in this population; 4. To evaluate four-month aerobic exercise and inspiratory muscle training on functional capacity, pulmonary function, and autonomic control in patients after Fontan operation and compare to the group with no exercise training.

Methods: All subjects were submitted to cardiovascular, pulmonary, and skeletal muscle evaluation at baseline to perform a cross-sectional study comparing Fontan Patients (FP) with Healthy Controls (HC). In addition, the FP accepted to participate in the longitudinal clinical trial to evaluate exercise programs were randomized into three groups: Aerobic Exercise Training (AET), Inspiratory Muscle Training (IMT), and Non-exercise Training Group (NET, a control group). All patient groups (AET, IMT, NET) were reassessed after four months of training or under usual care.

Expected Outcomes: This study expects to demonstrate that impaired pulmonary function, altered neurovascular control, and reduced skeletal muscle could be an additional potential mechanism for reducing functional capacity in clinically stable Fontan patients. And this impairment could be diminished by exercise training, enhancing physical capacity, and exercise tolerance.

DETAILED DESCRIPTION:
All subjects were submitted to cardiovascular magnetic resonance, echocardiography, cardiopulmonary exercise test, complete lung function, catecholamine and B-type natriuretic peptide (BNP) plasmatic levels, microneurography, venous occlusion plethysmography, six-minute walk test, phosphorus magnetic resonance spectroscopy (31P MRS) and magnetic resonance imaging (MRI) of skeletal muscle and quality of life (QoL) using the Short Form Health Survey (SF36) in the baseline. Comparative analyzes of the different systems of the two groups were done as well as tests to identify the predictors of low functional capacity in Fontan groups (FG).

The evaluation was done at baseline in healthy subjects. And in the Fontan group at baseline and after four months of exercise training or usual care.

AET Protocol: Four-month supervised exercise training was performed in the hospital three times a week, 60-min exercise sessions (48 sessions in total). Each session consisted of 40min on a treadmill, 15 min of personal light resistance training (including chest press, squat, pull down, leg extension, shoulder press, calf raises, leg curl, and sit-ups), and 5min of cool down and stretching. The AET was individually prescribed according to their heart rate (HR) from maximal cardiopulmonary exercise testing (CPT), and patients exercised between the ventilatory threshold (VT) and respiratory compensation point (RCP). HR, systolic blood pressure, oxygen saturation, and exhaustion (i.e., Borg scale from 7 to 20) were monitored during the sessions. An exercise physiologist supervised all sessions. In the first 12 weeks, HR was maintained at T frequency. Between the 12th to 24thweek, there was a progressive increase in the effort, and HR was supported between AT and RCP. In the last 12 sessions of the program, HR was maintained close to RCP frequency.

IMT Protocol: Four months of exercise training were carried out daily, three sets of 30 repetitions using the POWERbreathe® device (POWERbreathe International Limited, Southam, UK), three sets of 30 repetitions. Maximal inspiratory pressure (MIP) measures were performed in all patients before the intervention, and patients exercised at 60% of individual MIP. Patients were instructed to inhale using diaphragm musculature, trying to expand the rib cage to avoid the use of accessory muscles, and breathing at a rate of 12 to 16 breaths/min. A nose clip was worn to ensure patients breathed exclusively through the training device. All patients had a supervised session of IMT with a physiotherapist once a week for the first two months and once every two weeks for the last two months. The load was adjusted during the supervised sessions. Patients were encouraged to maintain their habitual activities during the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Both gender, aged between 12 and 30 years
* Patients undergoing the Fontan operation with time postoperatively ≥5 years
* Clinically stable patients, no arrhythmia in the last electrocardiogram or clinical assessment
* Consent by the cardiologist
* Patients who voluntarily signed the consent form.

Exclusion Criteria:

* Patients with hypoplastic left heart syndrome
* Changes that reduce musculoskeletal walking skills
* Neurological sequelae, patients with associated genetic syndrome, disturbance cognitive or psychiatric
* Patients with a history of ventricular arrhythmias, cardio respiratory arrest, users of anti-arrhythmic drugs and / or underwent implantation of pacemaker
* Atrial arrhythmia requiring treatment in the last 6 months
* Patients with heart failure not controlled by medications and lung hypertension
* Patients with protein-losing enteropathy
* Severe hypoxemia (oxygen saturation <80% at rest)
* Symptomatic patients with a diagnosis of diaphragmatic paresis or paralysis postoperative patients, with or without plication
* Patients with moderate to severe asthma
* Patients who live outside the area of Sao Paulo

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Improvement exercise tolerance and physical capacity | Baseline and 4 months
  Change in parameters by cardiopulmonary exercise test; increase in lung volumes and capacities; improvement by neurovascular control and skeletical muscle metabolism

OTHER OUTCOMES:
Improvement in the functional capacity post exercise training program | baseline and 4 months
  Increase at least 20% cardiopulmonary exercise test parameters: VO2 peak, oxygen pulse and VE/VCO2 slope
Improvement in pulmonary function post physical exercise program | baseline and 4 months
  Achieve at least 80% of predicted values for age at pulmonary function testing: spirometry, plethysmography, carbon monoxide diffusion capacity and maximal inspiratory pressure
Change in autonomic function post exercise training program | baseline and 4 months
  Decrease bursts/min and bursts per 100 heart beats by at least 20% from baseline by directly measured by microneurography : direct muscle sympathetic nerve activity (MSNA)
Improvement in peripheral blood flow post exercise training program | baseline and 4 months
  Increase forearm blood flow in mL/min/100mL
Change in the plasma epinephrine level post exercise training program | baseline and 4 months
  Decrease of plasma epinephrine level from baseline
Change in muscle metabolism post exercise training program | baseline and 4 months
  Increase of the amplitudes of the phosphocreatine, inorganic phosphate and ATP from baseline by 31P-MRS: Quadriceps femoral 31P-MRS

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo B Jatene, MD,PhD, Study Chair — Heart Institute, University of Sao Paulo, Medical School; Aida LR Turquetto, PhD student, Principal Investigator — Heart Institute, University of Sao Paulo, Medical School
Locations (1):
- InCor Heart Institute, São Paulo, Brazil

REFERENCES:
- [Background] Ohuchi H, Ohashi H, Takasugi H, Yamada O, Yagihara T, Echigo S. Restrictive ventilatory impairment and arterial oxygenation characterize rest and exercise ventilation in patients after fontan operation. Pediatr Cardiol. 2004 Sep-Oct;25(5):513-21. doi: 10.1007/s00246-003-0652-7. Epub 2004 May 12. PMID 15136907
- [Background] Brassard P, Poirier P, Martin J, Noel M, Nadreau E, Houde C, Cloutier A, Perron J, Jobin J. Impact of exercise training on muscle function and ergoreflex in Fontan patients: a pilot study. Int J Cardiol. 2006 Feb 8;107(1):85-94. doi: 10.1016/j.ijcard.2005.02.038. Epub 2005 Jul 19. PMID 16046016
- [Background] Binotto MA, Maeda NY, Lopes AA. Altered endothelial function following the Fontan procedure. Cardiol Young. 2008 Feb;18(1):70-4. doi: 10.1017/S1047951107001680. Epub 2007 Dec 20. PMID 18093358
- [Background] Steier J, Kaul S, Seymour J, Jolley C, Rafferty G, Man W, Luo YM, Roughton M, Polkey MI, Moxham J. The value of multiple tests of respiratory muscle strength. Thorax. 2007 Nov;62(11):975-80. doi: 10.1136/thx.2006.072884. Epub 2007 Jun 8. PMID 17557772
- [Background] Anderson PA, Sleeper LA, Mahony L, Colan SD, Atz AM, Breitbart RE, Gersony WM, Gallagher D, Geva T, Margossian R, McCrindle BW, Paridon S, Schwartz M, Stylianou M, Williams RV, Clark BJ 3rd; Pediatric Heart Network Investigators. Contemporary outcomes after the Fontan procedure: a Pediatric Heart Network multicenter study. J Am Coll Cardiol. 2008 Jul 8;52(2):85-98. doi: 10.1016/j.jacc.2008.01.074. PMID 18598886
- [Background] Trojnarska O, Gwizdala A, Katarzynski S, Katarzynska A, Szyszka A, Lanocha M, Grajek S, Kramer L. Evaluation of exercise capacity with cardiopulmonary exercise test and B-type natriuretic peptide in adults with congenital heart disease. Cardiol J. 2009;16(2):133-41. PMID 19387960
- [Background] d'Udekem Y, Cheung MM, Setyapranata S, Iyengar AJ, Kelly P, Buckland N, Grigg LE, Weintraub RG, Vance A, Brizard CP, Penny DJ. How good is a good Fontan? Quality of life and exercise capacity of Fontans without arrhythmias. Ann Thorac Surg. 2009 Dec;88(6):1961-9. doi: 10.1016/j.athoracsur.2009.07.079. PMID 19932269
- [Background] Greutmann M, Le TL, Tobler D, Biaggi P, Oechslin EN, Silversides CK, Granton JT. Generalised muscle weakness in young adults with congenital heart disease. Heart. 2011 Jul;97(14):1164-8. doi: 10.1136/hrt.2010.213579. Epub 2011 Jan 21. PMID 21258001
- [Result] Driscoll DJ, Durongpisitkul K. Exercise testing after the Fontan operation. Pediatr Cardiol. 1999 Jan-Feb;20(1):57-9; discussion 60. doi: 10.1007/s002469900397. No abstract available. PMID 9861079
- [Result] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Result] McCall R, Humphrey R. Exercise training in a young adult late after a fontan procedure to repair single ventricle physiology. J Cardiopulm Rehabil. 2001 Jul-Aug;21(4):227-30. doi: 10.1097/00008483-200107000-00007. No abstract available. PMID 11508184
- [Result] Minamisawa S, Nakazawa M, Momma K, Imai Y, Satomi G. Effect of aerobic training on exercise performance in patients after the Fontan operation. Am J Cardiol. 2001 Sep 15;88(6):695-8. doi: 10.1016/s0002-9149(01)01822-7. No abstract available. PMID 11564403
- [Result] Negrao CE, Rondon MU, Tinucci T, Alves MJ, Roveda F, Braga AM, Reis SF, Nastari L, Barretto AC, Krieger EM, Middlekauff HR. Abnormal neurovascular control during exercise is linked to heart failure severity. Am J Physiol Heart Circ Physiol. 2001 Mar;280(3):H1286-92. doi: 10.1152/ajpheart.2001.280.3.H1286. PMID 11179075
- [Result] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Result] Larsson ES, Eriksson BO, Sixt R. Decreased lung function and exercise capacity in Fontan patients. A long-term follow-up. Scand Cardiovasc J. 2003;37(1):58-63. doi: 10.1080/14017430310007045. PMID 12745804
- [Result] Inai K, Saita Y, Takeda S, Nakazawa M, Kimura H. Skeletal muscle hemodynamics and endothelial function in patients after Fontan operation. Am J Cardiol. 2004 Mar 15;93(6):792-7. doi: 10.1016/j.amjcard.2003.11.062. PMID 15019898
- [Result] Rhodes J, Curran TJ, Camil L, Rabideau N, Fulton DR, Gauthier NS, Gauvreau K, Jenkins KJ. Impact of cardiac rehabilitation on the exercise function of children with serious congenital heart disease. Pediatrics. 2005 Dec;116(6):1339-45. doi: 10.1542/peds.2004-2697. PMID 16322156
- [Result] Opocher F, Varnier M, Sanders SP, Tosoni A, Zaccaria M, Stellin G, Milanesi O. Effects of aerobic exercise training in children after the Fontan operation. Am J Cardiol. 2005 Jan 1;95(1):150-2. doi: 10.1016/j.amjcard.2004.08.085. PMID 15619417
- [Result] Inai K, Nakanishi T, Nakazawa M. Clinical correlation and prognostic predictive value of neurohumoral factors in patients late after the Fontan operation. Am Heart J. 2005 Sep;150(3):588-94. doi: 10.1016/j.ahj.2004.10.030. PMID 16169346
- [Result] Moalla W, Maingourd Y, Gauthier R, Cahalin LP, Tabka Z, Ahmaidi S. Effect of exercise training on respiratory muscle oxygenation in children with congenital heart disease. Eur J Cardiovasc Prev Rehabil. 2006 Aug;13(4):604-11. doi: 10.1097/01.hjr.0000201515.59085.69. PMID 16874152
- [Result] Takken T, Hulzebos HJ, Blank AC, Tacken MH, Helders PJ, Strengers JL. Exercise prescription for patients with a Fontan circulation: current evidence and future directions. Neth Heart J. 2007;15(4):142-7. doi: 10.1007/BF03085970. PMID 17612674
- [Result] Pianosi PT, Johnson JN, Turchetta A, Johnson BD. Pulmonary function and ventilatory limitation to exercise in congenital heart disease. Congenit Heart Dis. 2009 Jan-Feb;4(1):2-11. doi: 10.1111/j.1747-0803.2008.00244.x. PMID 19207396
- [Result] Goldstein BH, Golbus JR, Sandelin AM, Warnke N, Gooding L, King KK, Donohue JE, Gurney JG, Goldberg CS, Rocchini AP, Charpie JR. Usefulness of peripheral vascular function to predict functional health status in patients with Fontan circulation. Am J Cardiol. 2011 Aug 1;108(3):428-34. doi: 10.1016/j.amjcard.2011.03.064. Epub 2011 May 19. PMID 21600541
- [Result] Lambert E, d'Udekem Y, Cheung M, Sari CI, Inman J, Ahimastos A, Eikelis N, Pathak A, King I, Grigg L, Schlaich M, Lambert G. Sympathetic and vascular dysfunction in adult patients with Fontan circulation. Int J Cardiol. 2013 Aug 20;167(4):1333-8. doi: 10.1016/j.ijcard.2012.04.015. Epub 2012 Apr 21. PMID 22525342
- [Result] Turquetto ALR, Caneo LF, Agostinho DR, Oliveira PA, Lopes MICS, Trevizan PF, Fernandes FLA, Binotto MA, Liberato G, Tavares GMP, Neirotti RA, Jatene MB. Impaired Pulmonary Function is an Additional Potential Mechanism for the Reduction of Functional Capacity in Clinically Stable Fontan Patients. Pediatr Cardiol. 2017 Jun;38(5):981-990. doi: 10.1007/s00246-017-1606-9. Epub 2017 May 12. PMID 28500413
- [Result] Turquetto ALR, Dos Santos MR, Sayegh ALC, de Souza FR, Agostinho DR, de Oliveira PA, Dos Santos YA, Liberato G, Binotto MA, Otaduy MCG, Negrao CE, Caneo LF, Jatene FB, Jatene MB. Blunted peripheral blood supply and underdeveloped skeletal muscle in Fontan patients: The impact on functional capacity. Int J Cardiol. 2018 Nov 15;271:54-59. doi: 10.1016/j.ijcard.2018.05.096. Epub 2018 May 25. PMID 29861103
- [Result] Turquetto ALR, Dos Santos MR, Agostinho DR, Sayegh ALC, de Souza FR, Amato LP, Barnabe MSR, de Oliveira PA, Liberato G, Binotto MA, Negrao CE, Caneo LF, Trindade E, Jatene FB, Jatene MB. Aerobic exercise and inspiratory muscle training increase functional capacity in patients with univentricular physiology after Fontan operation: A randomized controlled trial. Int J Cardiol. 2021 May 1;330:50-58. doi: 10.1016/j.ijcard.2021.01.058. Epub 2021 Feb 9. PMID 33571562
- [Derived] Williams CA, Wadey C, Pieles G, Stuart G, Taylor RS, Long L. Physical activity interventions for people with congenital heart disease. Cochrane Database Syst Rev. 2020 Oct 28;10(10):CD013400. doi: 10.1002/14651858.CD013400.pub2. PMID 33112424